CLINICAL TRIAL: NCT05842499
Title: Substrate abLatIon as Concomitant trEatment for Left Atrial Macroreentrant Tachycardia - SLICE LAMRT
Brief Title: Substrate abLatIon as Concomitant trEatment for Left Atrial Macroreentrant Tachycardia
Acronym: SLICE-LAMRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Daniel Rodríguez Muñoz, Principal Investigator, Hospital Universitario 12 de Octubre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLICE-LAMRT
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
Keywords: Atypical atrial flutter; Ablation; Pulmonary veins; Macroreentrant Tachycardia; Scar; Atypical flutter
MeSH Terms: conditions — Atrial Fibrillation; Cicatrix

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The double-blind status will be established for the patient and the person responsible for the follow-up and clinical evaluation, who will never know the arm to which the patient has been randomized.
  Logically, this randomization will be known to the operator who will carry out the intervention, which will be performed on the basis of two treatment schemes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Line set strategy (Experimental): Pulmonary vein isolation, roof line, posterior wall isolation (posterior box), anterior septal line and cavo-tricuspid isthmus.
  Interventions: Procedure: Line Set Strategy
- Conventional strategy (Active Comparator): Mapping and ablation of the present flutter and those that could be induced later until sinus rhythm is obtained.
  Interventions: Procedure: Conventional strategy

INTERVENTIONS:
Procedure: Line Set Strategy — Substrate-guided ablation procedure of atypical atrial flutter
  Arms: Line set strategy
Procedure: Conventional strategy — Electrical activation-guided ablation
  Arms: Conventional strategy

SUMMARY:
SLICE-LAMRT is a multicenter, prospective, randomized, double-blind trial that will be carried out in patients older than 18 years with atypical flutter suspected to be of left atrial origin. The aim of this trial is to evaluate the safety and superiority of a substrate-guided ablation procedure vs the conventional strategy guided by electrical activity.

The composite primary endpoint is time to first episode of sustained atrial arrhythmia in the absence of pharmacological antiarrhythmic treatment or new ablation.

DETAILED DESCRIPTION:
Left atrial macroreentrant tachycardias (LAMRT), also known as left atrial flutter, represent a small percentage of supraventricular arrhythmiass. These tachycardias occur due to reentrant circuits, that is, electrical activation that occurs around natural anatomical obstacles or scar areas.

Classically, by analogy with ventricular tachycardias, these tachycardias are approached by delimiting the circuit (locating the anatomical and functional obstacles), searching for critical areas for their maintenance (isthmuses, generally of slow conduction) and creating controlled lesions that interrupt these circuits (catheter ablation). This requires electromagnetic mapping systems and uses programmed stimulation techniques. This approach treats flutter(s) present at the time of ablation to prevent recurrence. However, it is not uncommon for these patients to develop new macroreentrant circuits during the subsequent clinical course, so the recurrence rate of atrial arrhythmias in this population is relatively high.

The goal of this trial is to determine whether substrate-guided ablation of atypical atrial flutter is superior to electrical activation-guided ablation in reducing the recurrence of atrial arrhythmias and increasing the time to first recurrence of atrial fibrillation, atrial flutter, or atrial tachycardia. The investigators hypothesize that ablation not only of inducible tachycardias during the ablation procedure, but guided by the substrate that is most often key to the maintenance of these tachycardias, is superior to conventional treatment in reducing associated clinical events.

ELIGIBILITY:
Inclusion Criteria:

* Atypical flutter with positive F wave in V1, suspected left atrial origin.
* Age ≥ 18 years
* Capacity to understand the nature of the study, legal ability and willingness to give informed consent.

Exclusion Criteria:

* Simultaneous participation in a different trial.
* Presence of congenital heart disease.
* Suspected flutter of right origin or related to atriotomy scar from previous cardiac surgery.
* NYHA IV functional class at the time of recruitment.
* Contraindication to chronic anticoagulation or allergy/intolerance to heparin.
* Uncontrolled hyperthyroidism.
* Life expectancy less than 18 months.
* Presence of heart disease that is expected to require surgery or heart transplantation within 18 months.
* Pregnancy or the prospect of it in the next 18 months.
* Left atrium without pathological substrate: area ≥ 4 cm2 of low voltages (<0.5 mV) in the left atrium.
* Severe fragility (Clinical Frailty Score ≥ 7).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint | 18 months
  Time to first episode of sustained atrial arrhythmia in the absence of pharmacological antiarrhythmic treatment or new ablation

SECONDARY OUTCOMES:
Major complications | First month
  Death, stroke/systemic embolism, tamponade, during the procedure and immediate post-procedure.
Proportion of patients without recurrence of atrial arrhythmia at 18 months | 18 months
  Maintainance of sinus rhythm by ablation, without requiring electrical cardioversion.
Procedure duration | In the procedure
  Procedure duration, radiofrequency time, left atrial time (from transseptal puncture to left atrial catheter removal), fluoroscopy time.
Unplanned cardiovascular hospitalisation | 18 months
  Unplanned cardiovascular hospitalisation
Unplanned hospitalization for any cause. | 18 months
  Unplanned hospitalization for any cause.
All-cause mortality | 18 months
  Mortality due to any cause
Cardiovascular mortality | 18 months
  Mortality due to cardiovascular causes

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Arribas Ynsaurriaga, MD, PhD, Study Chair — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No